CLINICAL TRIAL: NCT04322955
Title: Cyto-KIK; TRIAL (CYTO Reductive Surgery in Kidney Cancer Plus Immunotherapy (Nivolumab) and Targeted Kinase Inhibition (Cabozantinib)
Brief Title: CYTO Reductive Surgery in Kidney Cancer Plus Immunotherapy and Targeted Kinase Inhibition
Acronym: Cyto-KIK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mark Stein (Other)
Collaborators: Exelixis (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Mark Stein, Associate Professor of Medicine Division of Hematology/Oncology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAS6927
Record Dates: First submitted 2020-02-10; First posted 2020-03-26 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — cabozantinib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Initially patients enrolled on the study will be assigned to Cohort 1. Patients assigned to Cohort 1 will have the cabozantinib held for three weeks prior to removal of the kidney. A patient in cohort 1 will be evaluable for assessment of the cabozantinib washout interval ("evaluable patients") if they
  1. complete at least 10 of the 14 scheduled cabozantinib doses in the two week period prior to stopping cabozantinib AND
  2. have surgical resection of the primary tumor.
  In cohort 2, subjects will receive cabozantinib until 14 days prior to nephrectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with cabozantinib and nivolumab with nephrectomy (Experimental): All study participants will receive the same study medications, cabozantinib and nivolumab. The study drug, nivolumab, will be administered through an IV infusion every 4 weeks and cabozantinib will be administered orally daily. Initially participants will receive study treatment for 12 weeks. The cabozantinib will then be stopped prior to the nephrectomy. Initially patients enrolled on the study will be assigned to cohort 1.
  Patients who are assigned to cohort 1 will be treated with cabozantinib until 21 days prior to surgery. A patient in cohort 1 will be evaluable for assessment of the cabozantinib washout interval ("evaluable patients") if they
  1. complete at least 10 of the 14 scheduled cabozantinib doses in the two week period prior to stopping cabozantinib AND
  2. have surgical resection of the primary tumor.
  In cohort 2, subjects will receive cabozantinib until 14 days prior to nephrectomy.
  Interventions: Drug: Cabozantinib; Drug: Nivolumab; Procedure: Cytoreductive nephrectomy

INTERVENTIONS:
Drug: Cabozantinib — 2 x 20 mg capsules taken orally daily
  Other Names: XL184
Drug: Nivolumab — 480mg IV on first day of each 28-day cycle
  Other Names: BMS-936558
Procedure: Cytoreductive nephrectomy — Surgery removing as much tumor tissue as possible, possibly including surrounding tissues.

SUMMARY:
The purpose of this study is to determine if the use of immunotherapy nivolumab and the targeted therapy cabozantinib prior to removal of the kidney, will increase the number subjects who are without any visible kidney cancer in their body at some point during the course of treatment.

DETAILED DESCRIPTION:
People with metastatic kidney cancer are usually treated with medications to slow the growth of the cancer. In addition, people who still have the kidney where the cancer started may have the kidney removed during the course of treatment. This surgery is done in order to decrease the amount of tumor in the body. This surgery is referred to as a cytoreductive nephrectomy. In the current study, nivolumab, an immune checkpoint inhibitor, is being administered in combination with cabozantinib, a targeted therapy. The combination of nivolumab and cabozantinib is FDA approved for the treatment of metastatic kidney cancer. In this study, treatment consists of cabozantinib and nivolumab plus a cytoreductive nephrectomy. Eligible subjects, who have not received prior therapy for metastatic clear cell renal cell carcinoma, are treated with cabozantinib and nivolumab for approximately 3 months prior to undergoing cytoreductive nephrectomy. After nephrectomy, patients who are benefiting from treatment may resume cabozantinib and nivolumab. This study will help investigators to understand the immune effects of cabozantinib and nivoluamb in the kidney tumor and will provide information on the potential clinical benefit associated with cytoreductive nephrectomy in combination with cabozanitnib and nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information.
2. Age ≥ 18years at the time of consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 within 28 days prior to registration.
4. Radiographically consistent with metastatic renal cell carcinoma (with subsequent pathologic confirmation of renal cell carcinoma with a clear cell component) OR histological/ cytological evidence of metastatic renal cell carcinoma with a clear cell component
5. Measurable tumor in the kidney according to RECIST 1.1
6. No prior therapy for metastatic renal cell carcinoma
7. Demonstrate adequate organ function as defined in the protocol; all screening labs to be obtained within 14 days prior to registration.
8. Females of childbearing potential must have a negative serum pregnancy test during screening, within 14 days of Cycle 1 Day 1. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
9. Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 6 months after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
10. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

1. Patients who had previously undergone nephrectomy for renal cancer are excluded
2. Uncontrolled bleeding, hypertension, or cardiovascular disease.
3. Prior treatment with any therapy on the PD-1/PD-L1 axis or anti- CTLA-4 inhibitors
4. The subject has active brain metastases or epidural disease
5. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment.
6. The subject has prothrombin time (PT)/ International Normalized Ratio (INR) or partial thromboplastin time (PTT) test ≥1.3 x the laboratory upper limit of normal (ULN)
7. The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, thrombin or Factor Xa inhibitors. Aspirin (up to 325 mg/day), low-dose warfarin (≤1 mg/day), prophylactic and therapeutic low molecular weight heparin (LMWH) are permitted
8. Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
9. Hemoptysis of ≥0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
10. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
11. The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
12. Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment
13. Patients are excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study start
14. Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic, or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 14 days of the first dose of study treatment.
    * The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) >500 ms within 28 days before registration.
15. Severe active infection requiring systemic treatment within 28 days before the first dose of study treatment
16. Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
17. Major surgery (e.g., GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (e.g., simple excision, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
18. History of organ transplant
19. Concurrent uncompensated hypothyroidism
20. Unable to swallow tablets
21. Active infection requiring systemic therapy
22. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
23. Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least 2 years.
24. Active central nervous system (CNS) metastases
25. Treatment with any investigational drug within 28 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with a Complete Response | Up to 5 years after completion of treatment
  The percentage of participants with a complete response following treatment. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

SECONDARY OUTCOMES:
Median Size Reduction of the Primary Tumor | 12 weeks
  Median size reduction of the primary tumor after treatment for 12 weeks prior to nephrectomy will be determined using RECIST 1.1 criteria applied to the primary tumor.
Progression Free Survival (PFS) | Up to 5 years after completion of treatment
  PFS is defined as the time from the time of first treatment on study until disease's progression or death as a result of any cause.
Response Rate | Up to 5 years after completion of treatment
  Response rate will include confirmed complete response (CR) + confirmed partial response (PR) and will be determined as per RECIST1.1.
Overall Survival | Up to 5 years after completion of treatment
  Overall survival will be measured from the time of first treatment on study until death or last follow-up.
Surgical Outcomes | Up to 5 years after completion of treatment
  Surgical outcomes will be assessed by the Clavien-Dindo classification system, which ranks the severity of surgical complications. The scale consists of several grades (Grade I, II, IIIa, IIIb, IVa, IVb and V) from Grade I being of low severity outcome to Grade V being highest and worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mark N Stein, MD, Principal Investigator — Associate Professor of Medicine Division of Hematology/Oncology
Locations (4):
- United States (4):
  - The Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio